CLINICAL TRIAL: NCT06194279
Title: Analysis of Different Postoperative Analgesia Strategies Following Scoliosis Surgery: Retrospective Study
Brief Title: Analysis of Different Postoperative Analgesia Strategies Following Scoliosis Surgery
Acronym: SAPOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8961
Record Dates: First submitted 2023-12-15; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Idiopathic Scoliosis
Keywords: Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Idiopathic scoliosis surgery is a major surgery, causing significant post-operative pain which can have a significant impact, both for the patient and for society. Different analgesic strategies have emerged in recent years, within the framework of multimodal analgesia including systemic analgesics, but also axial or peripheral loco-regional anesthesia (LRA). These techniques are integrated into the recommendations of learned societies, aimed at optimizing the post-operative rehabilitation of patients.

If intrathecal morphine injection (ITM) and spinal erector block (ESPB) have already shown their effectiveness in reducing postoperative pain, the combination of these techniques can have a real benefit in major spinal surgery. , and has not yet been studied.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged > 15 years
* Patient who underwent scoliosis surgery by the spine surgery team at Hautepierre hospital between January 1, 2020 and June 30, 2023
* Patient or holder of parental authority not opposing the reuse of their data for scientific research purposes

Exclusion Criteria:

* Oral or written refusal of the patient (or the holder of parental authority) to reuse their data for scientific research purposes
* History of spinal surgery
* Level 3 analgesics at home
* Protection of justice, titular or curatorship

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient aged > 15 years who underwent scoliosis surgery by the spine surgery team at Hautepierre hospital between January 1, 2020 and June 30, 2023
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Morphine dose administered 24 hours post-operative | 24 hours post-operative
  The aim of this retrospective study is to compare the different analgesic strategies postoperatively after scoliosis surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie Réanimation Médecine Péri Opératoire - CHU de Strasbourg - France, Strasbourg, France